CLINICAL TRIAL: NCT01601340
Title: A Randomized, Placebo-controlled, Phase 2 Study of HQK-1001 in Sickle Cell Disease
Brief Title: Effects of HQK-1001 in Patients With Sickle Cell Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: HemaQuest Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HQP 1001-SCD-007
Record Dates: First submitted 2012-05-12; First posted 2012-05-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia; Sickle Cell Disorders; Hemoglobin S Disease; Sickling Disorder Due to Hemoglobin S
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — 2,2-dimethylbutyric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HQK-1001 (Active Comparator)
  Interventions: Drug: HQK-1001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HQK-1001 — HQK-1001 tablets, twice daily for 48 weeks
  Arms: HQK-1001
Drug: Placebo — Placebo tablets, twice daily for 48 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of HQK-1001 on Hb F in subjects with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 12 and 60 years of age
* Diagnosis of SCD, type Hb SS or Hb S-B0 Thalassemia
* At least 1 episode of SCD pain crisis, acute chest syndrome, other acute SCD complications, or leg ulcers in the 12 months prior to screening
* Not being treated with Hydroxyurea (HU); if HU treatment has been previously administered and then discontinued, at least 3 months must have elapsed since last dose of HU
* If subject has been transfused in the 3 months prior to screening, then Hb A level < 20% at screening
* Baseline Hb F level obtained within 14 days prior to randomization
* Able to swallow tablets
* Able and willing to give informed consent and/or assent
* If subject is a woman of child-bearing potential (WCBP), she must have a negative serum pregnancy test within 14 days of first dose of HQK-1001 and a negative urine pregnancy test prior to dosing on Day 1
* If a subject is a WCBP, she must agree to use an effective form of contraception starting at screening and for one month after HQK-1001 discontinuation
* Sexually active male subjects who have not had a vasectomy must agree to use latex condoms with WCBP partners or ensure that their partner(s) use an effective form of contraception starting at screening and for one month after HQK-1001 discontinuation.

Exclusion Criteria:

* Assigned to a regular transfusion program
* Use of erythropoiesis stimulating agents within 90 days prior to screening
* An SCD pain crisis or SCD-related acute complication within 3 weeks prior to randomization
* More than 5 SCD pain crisis or SCD-related acute complications within 12 months prior to screening
* Pulmonary hypertension requiring therapy
* ALT or AST > 3x ULN
* Serum creatinine > 1.5x ULN
* Serum amylase levels > 1.5x ULN
* Serum lipase level > 1.5x ULN
* A serious, concurrent illness that would limit ability to complete or comply with the study requirements
* An acute illness (e.g., febrile, GI, respiratory) within 72 hours prior to screening
* History of syncope, clinically significant dysrhythmias or resuscitation from sudden death due to SCD-related complication
* Symptomatic peptic ulcer, hiatus hernia, or gastroesophageal reflux disease (GERD)
* History of pancreatitis
* Chronic opiate use, which, in the view of the investigator, could confound evaluation of an investigational drug
* Current abuse of alcohol or drugs
* Use of another investigational agent within 4 weeks or 5 half-lives, whichever is longer, prior to screening
* Currently pregnant or breast feeding a child
* Known infection with HIV-1
* Infection with hepatitis B or hepatitis C, such that subjects are currently on anti-viral therapy or will be placed on therapy

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2012-07; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in % fetal hemoglobin | Day 1 through Week 48

SECONDARY OUTCOMES:
Incidence and number of SCD pain crises and SCD-related complications | Day 1 through Week 52
Subject reported daily pain scale scores and analgesic use | 7 consecutive days following clinic visits at Day 1, and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Change in FACIT Fatigue Scale results | Day 1 and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Safety measured by the frequency and severity of adverse events, and changes from baseline in vital signs, electrocardiogram (ECG) monitoring, and laboratory assessments | Day 1 through Week 52
HQK-1001 pharmacokinetic parameters | 1 hour prior to, and 2 hours following morning dose on Weeks 12, 24 and 48
  A subset of subjects (7) will undergo sampling for detailed analysis of pharmacokinetic parameters (AUC, Cmax) with samples taken pre-dose, and 1, 2, 4, 8, and 10 hours after the morning dose at Week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ghalie, MD, MBA, Study Director — HemaQuest Pharmaceuticals Inc.
Locations (18):
- United States (11):
  - University of South Alabama, Mobile, Alabama
  - Children's Hospital and Research Center - Oakland, Oakland, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Georgia Health Sciences University, Augusta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - New York Methodist Hospital, Brooklyn, New York
  - The Children's Hospital at Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Virginia Commonwealth Univeristy - Center on Health Disparities, Richmond, Virginia
- University Health Network Toronto General Hospital, Toronto, Ontario, Canada
- Egypt (2):
  - Abu El Reesh Pediatric University Hospital, Cairo
  - Ain Sham University Hospital, Cairo
- University of the West Indies, Mona, Kingston 7, Jamaica
- Lebanon (3):
  - American University of Beirut Medical Center, Beirut
  - Chronic Care Center, Beirut
  - Rafik Hariri University Hospital, Beirut

REFERENCES:
- [Derived] Reid ME, El Beshlawy A, Inati A, Kutlar A, Abboud MR, Haynes J Jr, Ward R, Sharon B, Taher AT, Smith W, Manwani D, Ghalie RG. A double-blind, placebo-controlled phase II study of the efficacy and safety of 2,2-dimethylbutyrate (HQK-1001), an oral fetal globin inducer, in sickle cell disease. Am J Hematol. 2014 Jul;89(7):709-13. doi: 10.1002/ajh.23725. Epub 2014 Apr 15. PMID 24677033